CLINICAL TRIAL: NCT00107107
Title: A Multicenter, Open-Label, Extension Study of the Long-Term Safety of Pramlintide in Subjects With Type 1 Diabetes Mellitus Completing Protocol 137-150
Brief Title: Study of the Long-Term Safety of Pramlintide in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 137-150E
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Amylin; pramlintide; Symlin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — pramlintide

ARMS (1):
- Pramlintide Acetate (Active Comparator): Pramlintide acetate injection is a clear, colorless, sterile solution for SC injection. It consists of pramlintide in sodium acetate buffer, pH 4.0, containing 43 mg/mL mannitol as an iso-osmolality modifier and 2.25 mg/mL metacresol as a preservative. The concentration of pramlintide injection to be used in this study is 0.6 mg/mL.
  Interventions: Drug: pramlintide acetate

INTERVENTIONS:
Drug: pramlintide acetate — Syringe vial and Pen-cartridge

SUMMARY:
This is a multicenter, open-label extension study designed to examine the long-term safety of pramlintide treatment in subjects with type 1 diabetes who have successfully completed treatment in the parent study 137-150.

ELIGIBILITY:
Inclusion Criteria:

* The subject has completed the full dosing period in Protocol 137-150.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2002-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To investigate the long term safety profile of pramlintide treatment in subjects with type 1 diabetes completing protocol 137-150. | participant will be followed for the duration of the study, an average of 6 months or until Pramlintide is commercially available
To examine the long-term effect of subcutaneously (SC) injected pramlintide on body weight | participant will be followed for the duration of the study, an average of 6 months or until Pramlintide is commercially available

SECONDARY OUTCOMES:
To examine the effects of long term pramlintide treatment on HbA1c in subjects with type 1 diabetes completing protocol 137-150. | participant will be followed for the duration of the study, an average of 6 months or until Pramlintide is commercially available

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (25):
- United States (25):
  - Research Site, Tempe, Arizona
  - Research Site, Concord, California
  - Research Site, Fresno, California
  - Research Site, San Diego, California
  - Research Site, San Mateo, California
  - Research Site, Santa Barbara, California
  - Research Site, Walnut Creek, California
  - Research Site, Aventura, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Butte, Montana
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Irving, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Renton, Washington

REFERENCES:
- [Derived] Kovatchev BP, Crean J, McCall A. Pramlintide reduces the risks associated with glucose variability in type 1 diabetes. Diabetes Technol Ther. 2008 Oct;10(5):391-6. doi: 10.1089/dia.2007.0295. PMID 18715216